CLINICAL TRIAL: NCT00733889
Title: Phase II, Multicentre, Uncontrolled Pilot Study to Evaluate Safety and Efficacy of the Combination of Cetuximab and Chemotherapy (Docetaxel, Cisplatin, 5-fluorouracil) as Neoadjuvant Therapy Followed Concomitant Chemoradiotherapy (Cisplatin) Plus Cetuximab in Patients With a Locoregional Esophageal Carcinoma
Brief Title: A Study to Evaluate the Combination of Cetuximab and Chemotherapy as Neoadjuvant Therapy Followed Concomitant Chemoradiotherapy Plus Cetuximab in Locoregional Esophageal Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Spanish Cooperative Group for the Treatment of Digestive Tumours (TTD) (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TTD-06-02; EudraCT number:2006-001880-42
Record Dates: First submitted 2008-08-12; First posted 2008-08-13 (Estimated); Last update posted 2013-02-20 (Estimated); Status verified 2013-02

CONDITIONS: Esophageal Carcinoma
Keywords: esophageal carcinoma; cetuximab; docetaxel; cisplatin; 5-fluorouracil
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Cetuximab; Drug Therapy; Docetaxel; Cisplatin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: cetuximab and chemotherapy (docetaxel, cisplatin, 5-fluorouracil)

INTERVENTIONS:
Drug: cetuximab and chemotherapy (docetaxel, cisplatin, 5-fluorouracil) — Neoadjuvant chemotherapy plus cetuximab:
  3 cycles of chemotherapy (Docetaxel: 75 mg/m2; day1; Cisplatin :75 mg/m2, day 1; 5-FU: 750 mg/m2; 24-hour infusion; day1-5) administered every 3 weeks, plus cetuximab (250 mg/m2; day 1, 8 and 15) Cetuximab will be maintained from the beginning of chemotherapy until the end of radiotherapy.
  Radio-chemotherapy plus cetuximab:
  The radiotherapy treatment: A dose of 50.4 Gy will be administered in 28 fractions of 1.8 Gy / day, 5 days a week (a total of 5.6 weeks).
  Cetuximab:250 mg/m2 and Cisplatin: 40 mg/m2, day 1, 8, 15, 22, 29 and 36

SUMMARY:
The purpose of the study is to determine efficacy ans safety of the combination of cetuximab and chemotherapy (docetaxel, cisplatin, 5-fluorouracil) as neoadjuvant therapy followed concomitant chemoradiotherapy (cisplatin) plus cetuximab in patients with a locoregional esophageal carcinoma

ELIGIBILITY:
Inclusion Criteria:

* Informed consent form signed before performing any of the study's specific procedures.
* Age > 18 and < 70.
* Karnofsky performance status > 70% upon inclusion in the study.
* Life expectancy of more than 3 months.
* Histologically confirmed diagnosis of squamous cell carcinoma or adenocarcinoma of the oesophagus or the gastroesophageal junction. The disease must be confined to the oesophagus or gastroesophageal junction and the perioesophageal region. There must be no tumor extension beyond 2 cm into the stomach.
* Stages II or III. The patients must have a T1N1M0 or T2-4; any N; M0. The only exception would be patients with stage IVA: an oesophageal carcinoma of the upper thoracic region with metastasis in cervical lymph nodes (M1a) and an oesophageal carcinoma of the lower thoracic region with metastasis in the celiac lymph nodes (M1a), providing the disease remains within the radiotherapy fields.
* Presence of a unidimensionally measurable and/or assessable lesion
* Neutrophils >1500/mm3, platelet count >150,000/mm3 and haemoglobin >10 g/dl.
* Adequate renal function: serum creatinine < 120 micromol/l (1.4 mg/dl); if the values are >120 micromol/l (1.4 mg/dl) creatinine clearance must be > 65 ml/min.
* Adequate liver function: total bilirubin <1 x NUL; aspartate aminotransferase (AST) and alanine aminotransferase (ALT) <2.5 x NUL; alkaline phosphatase (AP) < 5 x NUL. Patients with AST and/or ALT > 1.5 < 2.5 x NUL and AP > 1.5 x NUL < 5 x NUL are not eligible.
* Serum calcium <1.25 x normal upper limit (NUL).
* Adequate nutritional status: weight loss < 20% of regular weight and albumin > 35 g/l.
* Total oral and/or enteral intake should be at least 1700 calories/day.
* Use of an effective contraceptive method for patients of both sexes when there is a risk of conception and/or pregnancy.
* Availability of tumour tissue for immunohistochemical analysis of EGFR expression and other biological markers.

Exclusion Criteria:

* Patients with a tracheo-oesophageal fistula or direct invasion of the tracheal mucosa or a major bronchi are not eligible. Bronchoscopy (with biopsy and cytology if lesion is seen) is required in order to rule out a fistula and/or direct invasion if the primary tumour is < than 30 cm from the incisors. Bronchoscopy is also required when the primary tumour is shown to be at or above the carina by an imaging study.
* Prior thoracic radiotherapy and/or systemic chemotherapy and/or oesophageal surgery.
* Patients with multiple carcinoma of the oesophagus.
* Diagnosis of any other cancer in the previous 5 years with the exception of appropriately treated carcinoma in situ of the uterine cervix and/or basal cell carcinoma of the skin.
* Systemic, chronic and concomitant immune treatment, or anti-cancer hormone therapy.
* Other concomitant cancer treatments.
* Active infection (infection requiring intravenous antibiotics), including active tuberculosis and diagnosed HIV.
* Uncontrolled hypertension defined as systolic blood pressure > 180 mmHg and/or diastolic blood pressure > 130 mmHg at rest.
* Active, uncontrolled, gastric or duodenal peptic ulcer.
* Chronic obstructive pulmonary disease requiring hospitalisation in the 6 months prior to inclusion in the study.
* History of atrioventricular arrhythmia and/or cardiac failure and/or second or third degree heart block.
* Clinically significant coronary artery disease or history of myocardial infarction in the last 12 months .
* Peripheral neuropathy grade > 2 NCIC-CTG of any aetiology.
* Hearing disorder grade > 2 NCIC-CTG of any aetiology.
* Any other disease or medical disorder suggesting that the patient will not be able to complete the study.
* Any psychological disorder suggesting that the complete treatment will not be possible.
* Pregnancy (its absence must be confirmed by the serum HCG-betatest) or lactation.
* Known drug abuse (with the exception of the mild or moderate consumption of alcohol upon inclusion in the study).
* Known allergic reaction to any of the components in the study treatment.
* Prior treatment with monoclonal antibodies or other signal transduction inhibitors or EGFR-targeted treatment.
* Evidence of another cancer, with the exception of a carcinoma in situ of the uterine cervix and/or a basal cell carcinoma of the skin.
* Any experimental treatment in the 30 days prior to inclusion in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2006-12; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
• Complete clinical response rate and objective clinical response rate after the administration of 3 cycles of chemotherapy plus cetuximab and after induction chemotherapy followed by concomitant chemoradiotherapy plus cetuximab | 2006-2010

SECONDARY OUTCOMES:
• To determine the complete pathological response rate in the patients subject to radical surgery, according to the investigators' criteria and the policy of each centre. | 2006-2010
Adverse events | 2006-2010
• To study the locoregional control of the disease, the therapeutic failure patterns, specific disease-free survival, event-free survival, disease-specific survival and global survival | 2006-2012
• To determine EGFR expression in the tumour and attempt to correlate it with efficacy | 2006-2010

CONTACTS AND LOCATIONS:
Overall Officials: Josep Tabernero, MD; phD, Study Chair — Medical Oncology Department; Hospital Universitario Vall d'Hebrón; Barcelona; Jordi Giralt, MD; phD, Study Chair — Oncology Radiation Department; Hospital Universitario Vall d'Hebrón; Barcelona
Locations (1):
- Spanish Cooperative Group for Gastrointestinal Tumour Therapy, Madrid, Spain

REFERENCES:
- [Derived] Alsina M, Rivera F, Ramos FJ, Galan M, Lopez R, Garcia-Alfonso P, Ales-Martinez JE, Queralt B, Anton A, Carrato A, Gravalos C, Mendez-Vidal MJ, Lopez C, de Mena IR, Tabernero J, Giralt J, Aranda E; Spanish Cooperative Group for the Treatment of Digestive Tumors (TTD) and Grupo de Investigacion Clinica en Oncologia Radioterapica (GICOR). A phase II Study Evaluating Combined Neoadjuvant Cetuximab and Chemotherapy Followed by Chemoradiotherapy and Concomitant Cetuximab in Locoregional Oesophageal Cancer Patients. Target Oncol. 2018 Feb;13(1):69-78. doi: 10.1007/s11523-017-0536-z. PMID 29128908